CLINICAL TRIAL: NCT02757807
Title: Stress Management Using an App to Improve Response With PDE5 Inhibitors in Men With Erectile Dysfunction.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eco Fusion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2016-04-26; First posted 2016-05-02 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Utilization of Serenita for Relaxation (Experimental): Intervention is that Users continue to take their PDE-5 Inhibitor prior to sexual interaction and IN ADDITION Utilize the Serenita App daily and before any sexual encounters.
  Interventions: Behavioral: Utilization of Serenita for Relaxation

INTERVENTIONS:
Behavioral: Utilization of Serenita for Relaxation — Users to use Serenita daily and before sexual interaction in order to assess stress and reduce it

SUMMARY:
The aim of this study is to determine if patients with ED taking PDE5 inhibitors (e.g. Viagra, CIalis, Levitra, Stendra) and experiencing performance anxiety will benefit using a user-friendly stress reducing phone app, Serenita. The study is internet based with no office visits.

DETAILED DESCRIPTION:
The etiology of erectile dysfunction (ED) has been investigated in many studies. Most often, ED is proposed to have a multifactorial etiology, with organic and/or psychogenic causal factors hypothesized to affect erectile function. Numerous studies show that Deep and Slow Breathing (DSB) reduces stress and anxiety.

Since ED is multifactorial, many physicians rely solely on phosphodiesterase-5 (PDE-5) inhibitors to increase blood flow to the arteries to maintain an erection. Although it works in many patients, some patients can get overly anxious prior to sexual intercourse and not be able to produce or maintain an erection. While some patients may realize that DSB may improve their anxiety they don't know how to perform DSB properly. We hypothesize that by providing software interactivity on deep and slow breathing to this group of ED patients, may in turn help reduce their anxiety, thus, maximize the effect of PDE5 inhibitors. The app called "Serenita" for mobile phones, designed by Eco-Fusion will be utilized in this study. The app performs two functions: it detects stress and focus level and It guides the user through a personalized breathing exercise designed to reduce stress and increase focus. Breathing as a method to treat stress has three scientifically validated variations, the deep diaphragmatic breathing, used for centuries as part of Yoga which often refers as Yogic breathing, biofeedback breathing, a method in which the user sees in real-time how his breathing affects his stress level, and coherence breathing, a method that synchronizes breathing pace with heart rhythms. The technology embedded in Serenita app combines all three methods into a personalized guided breathing regimen. The app acquires data by turning the mobile phone's camera into a biomedical sensor which peers into a person's blood stream, obtaining heart rate, heart rate variability and breathing pace. Then the app processes the data obtained to assess user's stress and focus level.

This study will utilize 6 standardized questionnaires to assess changes in patients' responses while using the app:

* Erectile Performance Anxiety Index (EPAI), which will ask questions that assess anxiety about being able to achieve or maintain an erection during sexual activity.
* International Index of Erectile Function (IIEF), which will ask questions about sexual encounters for the past four weeks.
* Psychological and Interpersonal Relationship Scales (PAIRS), which will ask questions about sexual self-confidence, time concerns and spontaneity with sexual encounters.
* Self-Esteem and Relationship (SEAR), which will ask questions about sexual relationship, confidence, stress ad perceived stress and overall sexual relationship for the past four weeks.
* Sexual Encounter Profile (SEP), which will ask question about each sexual attempt.
* Global Assessment Question, which will ask question at end of study if this app has improved erectile function.

These questionnaires are conducted online for easy access and completion. There are no office visits.

Registration to the study could be done at: http://eepurl.com/b3DcP1

ELIGIBILITY:
Inclusion Criteria:

* Male ages 18-55 years old
* Persistent mild to moderate ED on PDE5 inhibitors (Viagra, Cialis, Levitra, Stendra)
* Understand English
* Owns smartphone using either iPhone or Android
* Able to understand the use of "Serenita" app
* Willing to use Serenita app before sexual attempt
* Willing to complete all study questionnaires Willing to perform sexual attempt for at least once a week until end of study.

Exclusion Criteria:

* On testosterone replacement therapy
* History of Peyronie's disease
* Significant cardiac history (uncontrolled hypertension, cardiac arrhythmia, coronary artery disease, coronary bypass surgery)
* Uncontrolled diabetes mellitus
* History of prostate cancer
* Poorly controlled, symptomatic, active medical problems (HIV, hepatitis, cancer, benign prostatic hypertrophy, alcohol or drug abuse, major depressive disorder)
* Neurological or psychiatric disorder that would compromise the patient's ability to give informed consent or adhere to the requirements of the protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Global Assessment Profile measured by a survey | 1 month
  If the treatment has improved their erectile function

SECONDARY OUTCOMES:
Index of Erectile Function measured by a survey | 1 month
  if the treatment has improved erectile function

CONTACTS AND LOCATIONS:
Locations (1):
- RMA, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Companys website — http://www.eco-fusion.com